CLINICAL TRIAL: NCT02861469
Title: Reasons of Transfer in Emergency Units of Patients in End of Life Situation.
Acronym: CACTUS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2015/246
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: End of Life; Palliative Care
Keywords: qualitative study, end of life, ethics, palliative care
MeSH Terms: conditions — Death

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Main carers: Individual semi-structured interviews
  Interventions: Other: Semi-structured interviews
- General practitioners: Individual semi-structured interviews
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — individual semi-structured interviews with general practitioners and family members

SUMMARY:
This qualitative study aimed to describe and understand the factors leading to the admission in emergency unit of patients coming from their home, in an end of life situation.

This study was conducted in the university hospital of Besançon, France. Semi-structured interviews were conducted with general practitioners and family members in order to understand the factors leading, from their points of view, to the admission in emergency unit whereas this hospitalization wasn't necessary.

ELIGIBILITY:
Inclusion Criteria:

* FOR PATIENTS :
* aged of 18 yo or more
* Admitted in the emergency unit of the university hospital of Besançon
* who died within the 3 days following their admission in the emergency unit
* who died of a chronic disease in terminal phase
* for whom therapeutic goals were only focused on comfort
* living at their home or at their family's home before their transfer in emergency unit
* accompanied by at least one main carer (family member or friend) and one general practitioner during the last weeks before death
* FOR MAIN CARERS :
* Family members or friends of the patient
* who were the main carers of the patient during his/her last weeks
* speaking easily in french
* who agreed for being interviewed and whom psychic and emotional state is compatible with a interview
* living within 80km from Besançon
* FOR GENERAL PRACTITIONERS :
* who were the main medical actor for the patient during his/her last weeks
* who agreed for being interviewed
* working within 80km from Besançon

Exclusion Criteria:

* FOR PATIENTS :
* Patients who expressed a wish to not die at home
* Patients who died because of any other medical event than predictable death following the terminal phase of a chronic disease
* minors
* FOR MAIN CARERS AND GENERAL PRACTITIONERS :
* refusal to participate to the interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients living at their home and admitted in the emergency unit of the university hospital of Besançon, who died within the 3 days following their admission in the emergency unit of a chronic disease in terminal phase.
  * General practitioners and main carers (family members or friends) of those patients.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Perceptions of general practitioners and family members toward the reasons of admission in emergency unit of patients coming from home in an end of life situation | day one
  individual semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Régis AUBRY, Pr, Principal Investigator — Centre Hospitalier Universitaire de Besancon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Detering KM, Hancock AD, Reade MC, Silvester W. The impact of advance care planning on end of life care in elderly patients: randomised controlled trial. BMJ. 2010 Mar 23;340:c1345. doi: 10.1136/bmj.c1345. PMID 20332506
- [Background] Pennec S, Gaymu J, Monnier A, Riou F, Aubry R, Pontone S, Cases C. [The places of death of people aged 80 and over in France]. Soins Gerontol. 2014 Nov-Dec;(110):12-5. French. PMID 25597063